CLINICAL TRIAL: NCT00415662
Title: Effect of Biomagnetic Therapy on Gonarthrosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: HO 07/02
Record Dates: First submitted 2006-12-22; First posted 2006-12-25 (Estimated); Last update posted 2006-12-25 (Estimated); Status verified 2006-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

INTERVENTIONS:
Device: Pulsed Signal Therapy (PST)

SUMMARY:
In order to assess the effectiveness of biomagnetic therapy (PST) in the treatment of gonarthrosis, we conducted a randomized, double blind controlled clinical trial comparing one group of patients treated with PST and a second group of patients treated with conventional physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* at least 35 years old
* local symptoms over a period of at least one-year
* persistent symptoms despite non steroidal anti-inflammatory drugs
* informed consent

Exclusion Criteria:

* operative treatment in the last six months
* intra-articular injection in the last four months
* rheumatic disease
* homolateral coxarthrosis
* malignant disorder
* body mass index greater than 33%
* pregnancy
* inability to understand the visual analog scale

Min Age: 35 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2002-06; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: G Gremion, MD, Principal Investigator — HOSR
Locations (1):
- HOSR, Lausanne, Switzerland